CLINICAL TRIAL: NCT05527899
Title: Zinc Intervention in Elderly for Prevention of Pneumonia
Acronym: ZIPP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R34HL153277 (NIH); R34HL153277 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Zinc Deficiency
MeSH Terms: interventions — gluconic acid

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized, double-blind, placebo-controlled trial (RCT) in elderly NH residents with low serum Zn levels to evaluate the efficacy of 1 y of Zn supplementation (dose to be determined during R34 planning grant) in the prevention of PNA. Eligible subjects will be randomly assigned to one of two groups: both groups will receive a capsule containing ½ Recommended Dietary Allowance (RDA) of all the essential micronutrients, including 5 mg of elemental Zn; the Zn-supplemented group's capsule will contain an additional mg Zn gluconate (total equiv. of dose to be determined during R34 grant). Suppl. duration will be 12 mo to account for seasonal variations in the incidence of PNA.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will conduct a double-blind, randomized, and controlled trial (RCT) in elderly NH residents with low serum Zn levels (< 70 μg/dL ) to evaluate the efficacy of 1 y of 30 or 60 mg/d Zn supplementation on serum and T cell Zn levels, and T cell number and function. There will be a placebo group. Neither participants, nor Investgators or Outcome Assessors will be aware of treatment group. Masking will be done over RedCap Software and participants will be assigned to groups A, B, or C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): ½ RDA of micronutrients including 5 mg/d Zn
  Interventions: Drug: Zinc gluconate
- Zinc 30 mg (Experimental): ½ RDA of micronutrients including 30 mg/d Zn
  Interventions: Drug: Zinc gluconate
- Zinc 60 mg (Experimental): ½ RDA of micronutrients including 60 mg/d Zn
  Interventions: Drug: Zinc gluconate

INTERVENTIONS:
Drug: Zinc gluconate — 30 and 60 mg/d of zinc gluconate

SUMMARY:
Pneumonia is a major public health problem for the elderly and is one of the leading causes of hospitalization and death for this population, particularly for elderly nursing home residents. This planning grants seeks to establish a safe and effective dose of zinc supplementation with the goal to conduct a larger randomized clinical trial to study the effect of zinc supplementation in nursing home elderly with low serum zinc levels on the risk, antibiotic use, and duration of sick days with pneumonia. This project has significant potential to positively impact the health and quality of life in the elderly and to reduce the economic costs associated with their care.

DETAILED DESCRIPTION:
Pneumonia (PNA) is a leading cause of death and a major public health problem in the elderly, particularly for nursing home (NH) residents. Thus, there is an urgent need for effective strategies to prevent PNA in elderly. An important predisposing factor that may account for the higher incidence of PNA in older adults is the age-associated decline in T cell function. Importantly, there are remarkable similarities between Zn deficiency and age-induced changes in T cells. The investigators have shown that 29% of NH residents have low serum Zn levels, which was associated with higher incidence and duration of PNA, and antibiotic use. Although our preliminary data strongly suggest that low serum Zn is an independent risk factor for PNA in the elderly, a controlled clinical trial is critically needed to determine the efficacy of Zn supplementation in PNA prevention in this population. The objective of the larger clinical trial that will pursue the studies proposed in this R34 is to determine the effects of Zn supplementation on PNA outcomes in NH elderly and to understand their mechanistic basis. The central hypothesis is that improving Zn status in NH elderly with low serum Zn will reduce the incidence and duration of PNA, and the frequency of antibiotic use, and that the effect of Zn is mediated mainly through the improvement of T cell function. The rationale for conducting the proposed clinical trial is to determine the value of Zn supplementation as an inexpensive, easily implemented intervention that would aid in the prevention of PNA in the elderly. In a previous study NH elderly with low serum Zn levels, who were supplemented with 30 mg/d of Zn and ½ RDA of essential micronutrients showed, on average, significantly improved serum Zn levels. However, only 58% of participant became serum Zn adequate. The investigators therefore hypothesize that either a higher dose or a longer duration of supplementation is required to achieve adequate serum Zn levels in all Zn deficient elderly. The rationale for conducting the proposed pilot study is to determine the most effective yet safe dose for Zn supplementation in NH residents to be used in the larger clinical trial described above. The Specific Aim of the proposed two-year, pilot study is to establish the optimal dose of supplemental Zn to achieve adequate Zn status, and improved T cell function in Zn deficient elderly. This will be accomplished by conducting a randomized, placebo-controlled, double-blind clinical trial to test the efficacy of supplementation with 30 or 60 mg/d of Zn for 12 months on serum and T cell Zn levels, T cell function, and adverse events. The findings of this proposal are scientifically essential, yet sufficient, to allow us to make definitive decisions that inform the final design of our planned clinical trial, which aims to establish the value of Zn supplementation as an inexpensive, easily implemented intervention that would aid in the prevention of PNA, limit the duration of PNA, and consequently reduce the need for antimicrobial therapy in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly males and females (≥65 years)
2. >6 mo life expectancy, as judged by physician
3. Willing to be randomized into study groups
4. Able to swallow pills
5. Not currently on antibiotics
6. If consuming RDA levels of supplement, willing to replace with our control supplement
7. Calcium, vitamin D, and iron supplements permitted
8. Willing to receive influenza vaccine
9. BMI>18 kg/m2 and albumin >3.0 g/dL

Exclusion Criteria:

1. Anticipated transfer or discharge within 3 months of enrollment
2. Bed- or room-bound continuously for previous 3 months
3. Presence of lung neoplastic diseases or other active neoplastic diseases requiring chemotherapy and/or immunosuppressive drugs (including ≤10 mg/day prednisone)
4. Naso-gastric or other tube feeding
5. Long-term (≥30 days) IV or urethral catheters
6. Presence of tracheostomy or chronically ventilator-dependent
7. Chronic prophylactic antibiotic treatment or long term antibiotics
8. Those with PEM defined as albumin <3.0 g/dl and BMI <18kg/m2, 10
9. Consumption of supplements containing more than the RDA level of nutrients known to affect the immune response, i.e. vitamins E, C, B6, selenium, Zn, or beta-carotene
10. Diagnosis of PNA or other infection at baseline will not exclude a subject, but will postpone enrollment to 4 wks after PNA symptoms have cleared.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Zn levels | 12 months
  serum and intracellular Zn levels

SECONDARY OUTCOMES:
T cell profile | 12 months
  Total T cells, helper T cells, and cytotoxic T cells in PBMC will be determined by measuring populations of CD3, CD4, and CD8 positive cells, respectively, using flow cytometry.
T cell proliferation | 12 months
  PBMC will be incubated in the presence of T cell mitogens Con A or PHA, or antibodies against CD3 (T cell receptor) and CD28 (T cell co-receptor) for 72 h. Cultures will be pulsed with 0.5 μCi [3H]-thymidine (Perkin Elmer) during the last 4 h of incubation and then harvested onto glass-fiber mats (Wallac) with a Perkin Elmer cell harvester (Perkin Elmer). Cell proliferation will be assessed by the amount of [3H]-thymidine incorporated into the DNA as determined with the liquid-scintillation counting with a Micro Beta 2 MicroPlate counter (Perkin Elmer).
side effects | 12 months
  number of side effects will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ortega EF, Wu D, Guo W, Meydani SN, Panda A. Study protocol for a zinc intervention in the elderly for prevention of pneumonia, a randomized, placebo-controlled, double-blind clinical pilot trial. Front Nutr. 2024 Feb 21;11:1356594. doi: 10.3389/fnut.2024.1356594. eCollection 2024. PMID 38450236